CLINICAL TRIAL: NCT06015958
Title: Colonisation Efficacy of Streptococcus Salivarius M18 Toothpaste
Brief Title: Probiotic Toothpaste to Assess Microbial Colonization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BLIS Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BLTCT2022/9
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Microbial Colonization
Keywords: probiotic toothpaste; Streptococcus salivarius M18; Microbial colonization; Oral Probiotic; Toothpaste
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the 2 groups for brushing teeth with a probiotic toothpaste containing different doses of Streptococcus salivarius M18 Study Group A: BLIS M18 Toothpaste (10 million Cfu/dose) (n = 10) Study Group B: BLIS M18 Toothpaste (1 Million Cfu/dose) (n = 10)
Who Masked: Participant
Masking Description: A staff member not part of the study group will be assigned to distribute blinded samples. The participant or the investigators will not be aware of the dose groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Streptococcus salivarius M18 toothpaste dose 1 (Active Comparator): Streptococcus salivarius M18 toothpaste containing 1 million cfu/g
  Interventions: Other: Streptococcus salivarius M18 toothpaste (1 million cfu)
- Active Comparator: Streptococcus salivarius M18 toothpaste dose 2 (Active Comparator): Streptococcus salivarius M18 toothpaste containing 10 million cfu/g
  Interventions: Other: Streptococcus salivarius M18 toothpaste (10 million cfu)

INTERVENTIONS:
Other: Streptococcus salivarius M18 toothpaste (1 million cfu) — Probiotics Streptococcus salivarius M18 toothpaste 1 million cfu/g
  In this study, a toothpaste formulation containing S. salivarius M18 will be evaluated for its potential for delivering the probiotic to the oral cavity.
  Arms: Active Comparator: Streptococcus salivarius M18 toothpaste dose 1
Other: Streptococcus salivarius M18 toothpaste (10 million cfu) — Probiotics Streptococcus salivarius M18 toothpaste 10 million cfu/g
  In this study, a toothpaste formulation containing S. salivarius M18 will be evaluated for its potential for delivering the probiotic to the oral cavity.
  Arms: Active Comparator: Streptococcus salivarius M18 toothpaste dose 2

SUMMARY:
The aim of this study is to evaluate the colonization efficacy of probiotic toothpastes in healthy adults

DETAILED DESCRIPTION:
This is a double blind randomized controlled study with no cross over to evaluate the colonization efficacy of toothpaste containing a commercially available probiotic bacterium Streptococcus salivarius M18.

Participants will be randomly assigned to one of 2 groups for brushing teeth with a probiotic toothpaste containing two different doses of Streptococcus salivarius M18 over a seven day period. Saliva samples will be collected at predetermined time points pre and post intervention. Colonization efficacy will be determined by enumerating the probiotic in the saliva samples using standard microbiological techniques.

ELIGIBILITY:
Inclusion Criteria:

* In general good health
* Practise good oral hygiene

Exclusion Criteria:-

* Have a history of autoimmune disease or are immunocompromised.
* Are on concurrent antibiotic therapy or regular antibiotic use within last 1 week
* History of allergy (e.g. dairy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-11-29 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Microbial colonization from baseline (Day 0) to 1 hour | 1 hour post intervention
  Study will determine the change in the microbial colonization efficacy of two different doses of S. salivarius M18 in a toothpaste format.
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 in a toothpaste format. The saliva Statistical analysis (e.g. ANOVA) will be carried out to compare the participants data from baseline to one hour after later across three different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel, GraphPad Prism).
Change in Microbial colonization from baseline (Day 0) to 8 hours | 8 hours post intervention
  Study will determine the change in the microbial colonization efficacy of three different doses of S. salivarius M18 in a toothpaste format.
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 in a toothpaste format. The saliva Statistical analysis (e.g. ANOVA) will be carried out to compare the participants data from baseline to one hour after later across three different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel, GraphPad Prism).
Change in Microbial colonization from baseline (Day 0) to 24 hours | 24 hours post intervention
  Study will determine the change in the microbial colonization efficacy of three different doses of S. salivarius M18 in a toothpaste format.
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 in a toothpaste format. The saliva Statistical analysis (e.g. ANOVA) will be carried out to compare the participants data from baseline to one hour after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel, GraphPad Prism).
Change in Microbial colonization from baseline (Day 0) to 8 hours post last dose | 8 hours after last dose following 7 days of daily brushing with probiotic toothpaste.
  Study will determine the change in the microbial colonization efficacy of two different doses of S. salivarius M18 in a toothpaste format.
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 in a toothpaste format. The saliva Statistical analysis (e.g. ANOVA) will be carried out to compare the participants data from baseline to one hour after later across three different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel, GraphPad Prism).

CONTACTS AND LOCATIONS:
Locations (1):
- Blis Technologies Ltd, Dunedin, Otago, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burton JP, Drummond BK, Chilcott CN, Tagg JR, Thomson WM, Hale JDF, Wescombe PA. Influence of the probiotic Streptococcus salivarius strain M18 on indices of dental health in children: a randomized double-blind, placebo-controlled trial. J Med Microbiol. 2013 Jun;62(Pt 6):875-884. doi: 10.1099/jmm.0.056663-0. Epub 2013 Feb 28. PMID 23449874
- [Background] Bardellini E, Amadori F, Gobbi E, Ferri A, Conti G, Majorana A. Does Streptococcus Salivarius Strain M18 Assumption Make Black Stains Disappear in Children? Oral Health Prev Dent. 2020 Apr 3;18(2):161-164. doi: 10.3290/j.ohpd.a43359. PMID 32099975
- [Background] Di Pierro F, Zanvit A, Nobili P, Risso P, Fornaini C. Cariogram outcome after 90 days of oral treatment with Streptococcus salivarius M18 in children at high risk for dental caries: results of a randomized, controlled study. Clin Cosmet Investig Dent. 2015 Oct 3;7:107-13. doi: 10.2147/CCIDE.S93066. eCollection 2015. PMID 26491371